CLINICAL TRIAL: NCT01954576
Title: A Phase II Study of the Optune System, Enhanced by Genomic Analysis to Identify the Genetic Signature of Response in the Treatment of Recurrent Glioblastoma Multiforme
Brief Title: NovoTTF Therapy in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual; Avastin refractory patients not feasible given treatment paradigm in these patients.
Sponsor: University of Florida (Other)
Collaborators: Washington University School of Medicine (Other); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500287; 09-27-2013 (Other: Washington U IRB); 201306042 (Other: Washington U); OCR14655 (Other: University of Florida)
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Glioblastoma; Brain Neoplasms
Keywords: bevacizumab-naïve recurrent GBM; bevacizumab-refractory GBM
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NovoTTF therapy (Experimental): Patients undergo NovoTFF therapy at least 18 hours daily for 6 months (bevacizumab-naive) or 4 months (bevacizumab-refractory). Treatment may continue for up to 2 years in patients experiencing CR, PR, or SD.
  Interventions: Device: NovoTTF-100A; Procedure: Quality-of-life assessment; Genetic: Laboratory biomarker analysis

INTERVENTIONS:
Device: NovoTTF-100A
Procedure: Quality-of-life assessment
Genetic: Laboratory biomarker analysis

SUMMARY:
This pilot phase II trial studies how well Novocure's Tumor Treating Electric Fields (NovoTTF) therapy works in treating patients with recurrent glioblastoma multiforme. NovoTTF therapy uses a low intensity electric current to kill tumor cells. NovoTTF therapy may be effective treatment for brain cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM (WHO grade IV); rare GBM variants (e.g. gliosarcoma, giant cell GBM, small cell GBM, GBM with oligodendroglioma features, GBM with PNET features) are allowed. Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of GBM is made.
* Received radiotherapy of at least 45 Gy and temozolomide chemotherapy as initial treatment for GBM.
* Unequivocal evidence of recurrent or progressive GBM before or after bevacizumab treatment first based on radiographic appearances then confirmed by histologic confirmation through biopsy or resection.
* Prior treatment with Gliadel wafer is allowed if it has been at least 3 months from placement.
* There must be an interval of at least 12 weeks from the completion of radiotherapy to start of device treatment. When the interval is less than 12 weeks from the completion of radiotherapy, the histological confirmation of progression must be unequivocal per RANO criteria. The use of PET scan, perfusion imaging, and MRspectroscopy to differentiate between true early progression and pseudoprogression prior to biopsy or resection of probable recurrent tumor is per standard of care.
* At least 22 years of age.
* Karnofsky performance status of at least 60%.
* Life expectancy of at least 3 months.
* Planned biopsy or resection of recurrent tumor for therapeutic and/or diagnostic purpose, and with adequate bone marrow, hepatic, cardiac, and renal function to undergo this planned procedure.
* For patients who have undergone or will undergo stereotactic biopsy of recurrent or progressive tumor, a post-operative MRI is not required, provided that the pre-biopsy MRI is within 21 days of registration. If the preoperative scan is more than 21 days before registration, the scan needs to be repeated. If the steroid dose is increased more than 50% between the date of biopsy and registration, a new baseline MRI is required on a stable or decreasing steroid dosage for at least 3 days even if the previous MRI was within 21 days of registration.
* For patients who have undergone or will undergo open resection of recurrent or progressive tumor, residual disease following resection is not mandated for eligibility into the study. To best assess the extent of residual disease post-resection, a MRI scan should be done no later than 96 hours in the immediate post-resection period and within 21 days prior to registration. If the 96-hour scan is more than 21 days before registration, the scan needs to be repeated. If the steroid dose is increased more than 50% between the date of imaging and registration, a new baseline MRI is required on a stable or decreasing steroid dosage for at least 3 days.
* Planned treatment with NovoTTF Therapy alone per FDA-approved indication. NovoTTF Therapy must start within 14 days of registration, but not less than 7 days or more than 21 days from stereotactic biopsy (if applicable) and not less than 21 days or more than 42 days from open resection (if applicable).
* Availability of tissue from the initial diagnosis and the recurrent tumor that is estimated to be of sufficient quality and quantity for both genomic DNA and total RNA isolation; preferably some of the tissue would be snap frozen for high quality RNA preparation.
* Because the genetic analyses described in Section 8.0 will be performed under HRPO# 201111001 ("Analysis of Histological, Genomic, Molecular, and Clinical Factors in CNS Cancer: the Neuro-Oncology Group"), for patients enrolling in this trial at WUSM, it is required that WUSM patients must also enroll in HRPO# 201111001. The genetic analyses for UF patients will take place at WUSM under the auspices of this protocol.
* Recovery from the toxic effects of prior therapy to not more than grade 1 or >3 weeks from prior therapy to registration, whichever is later.
* Patients must agree to forgo any other treatments, including but not limited to cytotoxic or biologic chemotherapies, that are intended to treat the recurrent GBM while receiving treatment with NovoTTF Therapy.
* Participants of childbearing age must use effective contraception.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Any other malignancy that required active chemotherapy within the previous 12 months prior to registration and the disease is not currently progressing and/or metastatic. The exception is basal cell or squamous cell carcinoma of the skin, which were treated with local resection only or carcinoma in situ of the cervix.
* Unable to undergo brain MRI due to medical or personal reasons.
* Bevacizumab-naïve patients: These patients may not have more than one prior relapse not counting the current relapse being treated by this protocol and must have received at least one prior chemotherapy regimen, which must have included temozolomide.
* Bevacizumab-refractory patients: These patients may not have more than 2 prior relapses not counting the current relapse being treated by this protocol and must have received multiple chemotherapy regimens, including a temozolomide regimen and a bevacizumab regimen.
* Currently receiving any other investigational agents that are intended as treatments of recurrent GBM.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or severe heart problems, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding.
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, vagus nerve stimulator, and other implanted electronic devices in the brain or the spinal cord.
* Infra-tentorial tumor.
* History of hypersensitivity to hydrogel.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
ORR (CR + PR + SD) (bevacizumab-naive) | 6 months
  Response and progression evaluated using Response Assessment in Neuro-Oncology (RANO). Response is evaluated with the use of MRI every 8 weeks. A Fisher's exact test with two-sided 0.05 and 80% power will be used.
ORR (CR + PR + SD) (bevacizumab-refractory) | 4 months
  Response and progression evaluated using Response Assessment in Neuro-Oncology (RANO). Response is evaluated with the use of MRI every 8 weeks. A Fisher's exact test with two-sided 0.05 and 80% power will be used.

SECONDARY OUTCOMES:
Genetic signature of response (CR + PR + SD) | up to 6 months
  Genetic analysis will be performed on the primary tumor tissue and tissue at the time of recurrence. Genomic DNA will be extracted from patients' tumor samples and paired blood samples.
Genetic signature of response (CR + PR) and SD | Up to 6 months
  Genetic analysis will be performed on the primary tumor tissue and tissue at the time of recurrence. Genomic DNA will be extracted from patients' tumor samples and paired blood samples.
Progression-free survival in bevacizumab-naïve and bevacizumab-refractory glioblastoma patients | Assessed up to 2 years
  Defined as start of treatment to time of progression or death, whichever occurs first. Will be estimated by Kaplan-Meier curves.
Quality of Life | Up to 30 days post-treatment
  Assessed using the Karnofsky performance status and the mini-mental state examination.

CONTACTS AND LOCATIONS:
Overall Officials: David Tran, M.D., Ph.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu